CLINICAL TRIAL: NCT01510145
Title: Multi-Center Study Comparing Efficacy and Tolerability of TRAVATAN® BAK-free (0.004% Travoprost) in Patients Previously on Latanoprost Ophthalmic Solution 0.005% Monotherapy
Brief Title: Efficacy of Changing to TRAVATAN® From Prior Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-10-300
Record Dates: First submitted 2012-01-11; First posted 2012-01-13 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Open-angle glaucoma; Ocular hypertension; Hypertension; Eye Diseases; Vascular Diseases; Cardiovascular Diseases; Travoprost; Antihypertensive Agents; Cardiovascular Agents; Therapeutic Uses; Pharmacologic Actions
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension; Eye Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRAVATAN® BAK-free (Experimental): Travoprost 0.004% BAK-free, 1 drop self-administered to the study eye(s) once daily, every evening at around 8:00 pm, for 12 weeks.
  Interventions: Drug: Travoprost 0.004% BAK-free

INTERVENTIONS:
Drug: Travoprost 0.004% BAK-free — Containing Polyquad (PQ) preservative
  Other Names: TRAVATAN® BAK-free

SUMMARY:
The purpose of this study was to assess the efficacy and tolerability of TRAVATAN® solution without BAK (benzalkonium chloride) after changing from prior latanoprost 0.005% ophthalmic solution monotherapy in subjects with open-angle glaucoma or ocular hypertension due to tolerability issues.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension or open-angle glaucoma in at least one eye;
* On latanoprost ophthalmic solution 0.005% monotherapy (including BAK-containing generics) for at least 4 weeks prior to the Screening Visit, but would benefit from a switch to TRAVATAN® BAK-free because of tolerability issues, in the opinion of the investigator;
* Intraocular pressure (IOP) <30 millimeters of mercury (mmHg) in both eyes while on latanoprost ophthalmic solution 0.005% monotherapy;
* IOP considered to be safe (in the opinion of the investigator), in both eyes, in such a way that assured clinical stability of vision and the optic nerve throughout the study period;
* Willing to discontinue the use of all other ocular hypotensive medications prior to receiving the study medication for the entire course of the study;
* Able to follow instructions and willing and able to attend all study visits;
* Best corrected Snellen visual acuity of 6/60 (20/200; 1.0 LogMAR) or better in each eye;
* Must sign an informed consent form;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity, or poor tolerance to any component of the preparations to be used in this study deemed clinically significant in the opinion of the Principal Investigator;
* Any abnormality preventing reliable applanation tonometry in either eye;
* Corneal dystrophies in either eye;
* Concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye;
* Any clinically significant, serious, or severe medical condition;
* Use of any systemic medications known to affect IOP which have not been on a stable course for at least 7 days prior to the Screening Visit or an anticipated change in the dosage during the course of the study;
* Severe dry eye or keratoconjunctivitis sicca which has been or is currently being treated with the use of punctal plugs, punctal cautery, Restasis®, or topical ocular corticosteroids;
* Intraocular conventional surgery or laser surgery in either eye less than 3 months prior to the Screening Visit;
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment;
* Progressive retinal or optic nerve disease from any cause;
* Women who are pregnant, lactating, or not using reliable means of birth control;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana S. Bonadia, Study Director — Alcon Research

REFERENCES:
- [Derived] Lopes JF, Hubatsch DA, Amaris P. Effect of benzalkonium chloride-free travoprost on intraocular pressure and ocular surface symptoms in patients with glaucoma previously on latanoprost: an open-label study. BMC Ophthalmol. 2015 Nov 12;15:166. doi: 10.1186/s12886-015-0151-7. PMID 26563363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 4 study centers located in Argentina, 4 study centers located in Chile, and 2 study centers located in Colombia.
Pre-assignment Details: This reporting group includes all enrolled patients (191).
Groups:
- TRAVATAN® BAK-free: Travoprost 0.004%, 1 drop self-administered to the study eye(s) once daily, every evening at around 8:00 pm, for 12 weeks.
Period: Overall Study
Arm/Group | TRAVATAN® BAK-free
Started | 191
Completed | 173
Not Completed | 18
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 6
Not completed — Relative reported subject withdrew | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled patients.
Arm/Group | TRAVATAN® BAK-free
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) at 12 Weeks From Prior Therapy (Baseline)
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater amount of improvement. One eye was chosen as the study eye, and only data from the study eye were used for the efficacy analysis.
Time Frame: Baseline, Week 12
Population: This analysis population includes all patients who instilled at least one drop of study product and who had primary endpoints measures available for at least one on-therapy study visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TRAVATAN® BAK-free
Number analyzed (Participants) | 191
mmHg
  Baseline | 14.8 (3.4)
  Change from baseline at Week 12 | -1.09 (2.96)

2. Secondary Outcome: Percentage of Subjects Who Reach Target IOP (≤18 mmHg)
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye was chosen as the study eye, and only data from the study eye were used for the efficacy analysis.
Time Frame: Week 12
Population: This anaylysis population includes all subjects who instilled at least one drop of study product and who had primary endpoints measures available for at least one on-therapy study visit.
Measure: Number; unit: percentage of patients
Arm/Group | TRAVATAN® BAK-free
Number analyzed (Participants) | 191
percentage of patients | 93.3

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (1 year, 3 months). This analysis group includes all patients who instilled at least one drop of test article.
Description: AE data were collected and reported in the eCRF at each visit from time of first drug instillation to Week 12.
Arm/Group | TRAVATAN® BAK-free
Serious Adverse Events (participants affected / at risk) | 0/191
Other Adverse Events (participants affected / at risk) | 0/191

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.